CLINICAL TRIAL: NCT03164408
Title: High Early Post-operative Complication Rate After Elective Aseptic Orthopedic Implant Removal of Upper and Lower Limb
Brief Title: Orthopaedic Implant Removal
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Arnold J Suda, MD, PhD, Senior Consultant Orthopaedic and Trauma Surgeon, Universitätsmedizin Mannheim
Other Study IDs: 2017/01SUA
Record Dates: First submitted 2017-05-21; First posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Implant Complication; Complication, Postoperative; Implant Site Infection
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Orthopaedic Implant Removal

SUMMARY:
The necessity of orthopedic implant removal is under intense discussion and even if it is performed as an elective procedure, the risk of complications is present.

Aim of the study is to identify parameters responsible for an increased risk of early post-operative complications after elective aseptic orthopedic implant removal.

ELIGIBILITY:
Inclusion Criteria:

Elective aseptic orthopaedic Implant removal

Exclusion Criteria:

Arthroplasty present infection

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: all patients in between scheduled period of time ( 2 years)
Sampling Method: Probability Sample
Enrollment: 1545 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2017-04-05 (Actual)

PRIMARY OUTCOMES:
Complications after implant Removal | 4 weeks postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Arnold J Suda, MD, PhD, Principal Investigator — University Medical Center Mannheim

IPD SHARING:
Plan to Share IPD: No